CLINICAL TRIAL: NCT04976205
Title: Artificial Intelligence Algorithms to Automate the Total Marrow (Lymph-node) Irradiation by VMAT Optimization Using WB-CT/MRI and Synthetic WB-CT - The AuToMI Project
Brief Title: AI Algorithms to Automate the TMI by VMAT Optimization Using WB-CT/MRI and Synthetic WB-CT - The AuToMI Project
Acronym: AuToMI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2928
Record Dates: First submitted 2021-06-30; First posted 2021-07-26 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Hematological Disease
MeSH Terms: conditions — Hematologic Diseases | interventions — Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TMI/TMLI (Experimental): The standard planning optimization for TMI/TMLI preview a two-free-breathing-CT scan without contrast will be performed for simulation at day -15(-10) to the BMT. The same day a WB-MRI will be acquired for lymph-nodes delineation. WB-MRI scans will be performed using a 1.5T MR scanner. The two CT will be co-registered to the WB-MRI.
  CTV will be manually defined as the bones excluding mandible and hands (CTVBones), the spleen (CTVSpleen), and lymph nodes (CTVLN) using both MRI and CT images. The day -3 (4) to the BMT, further two-CT series will be acquired and co-registered to the first CTs for dose verification. Pre-treatment quality assurance (QA) will be performed the day before the treatment using the standard internal procedure.
  The treatment will be performed the day before the BMT.
  Interventions: Radiation: Total Marrow (Lymph-node) Irradiation

INTERVENTIONS:
Radiation: Total Marrow (Lymph-node) Irradiation — To the standard procedure for TMI/TMLI target definition, based on simulation WB-CT acquired 10/15 days before BMT, we acquire: WB- magnetic resonance imaging (MRI) the same day of the simulation WB-CT. A verification WB-CT will be performed 3/4 days before the delivery. Plans will be optimized with Volumetric Modulated Arc Therapy (VMAT) technique.

SUMMARY:
Total Body Irradiation (TBI) was shown to help in providing immunosuppression that facilitates the donor transplant acceptance. Randomized trials demonstrated that conditioning regimens to bone marrow transplantation (BMT) including TBI have produced better survival rates than chemo-only regimens. The TBI target is represented by the whole BM, and eventually the whole lymphatic system, liver, spleen. The increased life expectancy revealed the occurrence of important toxicities because of full doses received by organs at risk (OARs) and this limited the use of TBI. Many groups have explored the possibility of sophisticated techniques for reducing the dose to healthy tissues while increasing the dose to the BM. These newer approaches aim to generate total marrow (lymph-node) irradiation (TMI/TMLI), sparing as much as possible non-skeletal and non-lymphoid structures.

Actually, the time required to optimize a TMI/TMLI plan is 10 days. Therefore, the simulation Computed Tomography (CT) is performed many days before the BMT. Furthermore, the lymph-nodes are defined only on CT images.

DETAILED DESCRIPTION:
Total Body Irradiation (TBI) was shown to help in providing immunosuppression that facilitates the donor transplant acceptance. Moreover, TBI plays a role in the annihilation of malignant cells, and may also deplete normal hematopoietic stem cells, thus helping the donor marrow cells to repopulate the bone marrow (BM). Randomized trials demonstrated that conditioning regimens to BMT including TBI have produced better survival rates than chemo-only regimens.

The TBI target is represented by the whole BM, and eventually the whole lymphatic system, liver, spleen. Usually, a very simple geometry is adopted, with patient positioned on a dedicated couch at 3-4 meters away from the linear accelerator to fully cover the target with a single beam, avoiding field junctions.

The increased life expectancy revealed the occurrence of important toxicities because of full doses received by organs at risk (OARs) and this limited the use of TBI as stated by the 2018 ILGROG guidelines. Many groups have, therefore, explored the possibility of sophisticated techniques for reducing the dose to healthy tissues while increasing the dose to the BM. These newer approaches aim to generate total marrow (lymph-node) irradiation (TMI/TMLI), sparing as much as possible non-skeletal and non-lymphoid structures.

Preliminary clinical data on phase I/II trials support the use of TMI/TMLI as part of conditioning for BMT for relapsed-refractory acute leukemia patients and multiple myeloma. However, TMI/TMLI adoption is still very limited to few skilled hospitals due to the extreme difficulty in the planning that needs many days.

The evaluation of TMI/TMLI with Volumetric Modulated Arc Therapy (VMAT) was started in our institute in 2009 and we treated around 90 patients in 10 years.

VMAT-TMI/TMLI requires multiple arcs from isocenters with different positions to fully include the patient length. Therefore, many field junctions between arcs with different isocenters should be managed. Furthermore, the CT length does not allow to acquire the patient in a single CT scan. Two CT series must be acquired and co-registered.

Actually, the time required to optimize a TMI/TMLI plan is 10 days. Therefore, the simulation Computed Tomography (CT) is performed many days before the BMT. Furthermore, the lymph-nodes are defined only on CT images.

Deep learning (DL) artificial intelligence (AI) algorithms in medical imaging and RT are rapidly expanding. DL focused on lesion detection and classification by features extraction. Image segmentations using fully convolutional network (FCN), holistically nested network (HNN) or other customized network architectures were implemented in many regions.

Over the past decades, the use of magnetic resonance imaging (MRI) to support RT has increased. MRI provides excellent soft-tissue imaging that could improve the target definition. The lymph-nodes contouring, based on MRI, will result in smaller target, enabling a better sparing of healthy tissues. Moreover, MRI significantly reduces inter/intra-observer contouring variability. At this aim, new generation MRI consoles with larger bore size, flat tabletops and dedicated imaging protocols with reduced image distortion to <1 mm were developed. Moreover, newly developed gradient-echo 3D sequences, and dedicated coils, can be used for producing a whole body WB-MRI acquisition in a few minutes. Furthermore, synthetic CT from MRI was proposed and implemented in some regions (i.e. brain and prostate) to substitute the CT for providing electron density information for dose planning calculation.

ELIGIBILITY:
Inclusion Criteria:

* Written, signed informed consent
* Adult patients aged ≥18 years
* Diagnosis of Hematological disease
* Eligibility for allogeneic stem cell transplantation as center guidelines
* TMI/TLI as part of the conditioning regimen

Exclusion Criteria:

- Conditioning regimen including only chemotherapeutic agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-06-15 (Actual); Primary Completion 2025-08-08 (Actual); Study Completion 2025-08-08 (Actual)

PRIMARY OUTCOMES:
Reduction of Lymph nodes target volume thanks to WB-MRI | 3 years
  The PTV_LN volumes generated on the Simulation WB-MRI and on the Simulation WB-CT will be compared.

SECONDARY OUTCOMES:
Doses calcuated on CT performed at day -3 (4) to the BMT | 3 years
  To evaluate the dosimetric changes that occurs in the days between the simulation and the delivery.
  The RT plan is defined on a simulation CT perfomed at -15 days. A second CT is performed at day -3 (4) to the BMT. The RT plan is recalculated on the second CT. The PTV volume receiving 95% of doses will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Humanitas Research Center, Rozzano, Milano, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Dei D, Lambri N, Sopranzi C, Galdieri C, Franzese C, Scorsetti M, Mancosu P. Impact of reduced interval from simulation CT to treatment delivery on dosimetric and positioning accuracy for total marrow lymph-node irradiation. Strahlenther Onkol. 2025 Jun 13. doi: 10.1007/s00066-025-02415-x. Online ahead of print. PMID 40512423